CLINICAL TRIAL: NCT02702817
Title: Investigations of Naproxen Treatment Effects in Pre-clinical Alzheimer's Disease (INTREPAD)
Brief Title: Randomized Trial of Low-dose Naproxen in Cognitively Intact Persons at Risk of Alzheimer's Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: McGill University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, John C. S. Breitner, Director, Centre for Studies on Prevention of Alzheimer's Disease, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INTREPAD
Record Dates: First submitted 2015-12-19; First posted 2016-03-09 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer Disease; Cognitive Decline Due to Alzheimer Disease; Mild Cognitive Impairment Due to Alzheimer Disease
Keywords: Alzheimer's disease, biomarkers, cognitive decline, pre-clinical
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Naproxen; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- naproxen (Active Comparator): naproxen sodium tablets 220 mg twice daily for two years
  Interventions: Drug: Naproxen
- placebo (Placebo Comparator): tablets identical in appearance to naproxen tablets twice daily for two years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen — pale blue oval tablets
  Other Names: Naprosyn, Anaprox, Aleve
  Arms: naproxen
Drug: Placebo — pale blue oval tablets with no active ingredients, identical in appearance to naproxen intervention
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
Two-year double-masked trial of over-the-counter dosage of naproxen sodium vs placebo in 200 cognitively normal participants with a parental or multiplex first-degree family history Alzheimer's disease (AD) dementia. Primary outcomes are decline in cognitive function and slope of change in a summary Alzheimer Progression Score derived from serial assessment of neuroimaging, biochemical, and sensori-neural biomarker indicators of pre-clinical disease -- all believed likely to reflect progress of preclinical AD in this high risk cohort. Approximately 2/3 of participants have volunteered also for serial lumbar punctures for analysis of cerebrospinal fluid. A two-year off-treatment delayed-washout phase is planned to examine sustained treatment effects and evidence of disease modification.

DETAILED DESCRIPTION:
The trial enrolled 195 cognitively normal persons aged 60+ with either a parental history of AD or a history of two or more affected first-degree relatives. Persons aged 55-59 were admitted if their current age was <= 15 years younger than AD onset in their index relative. Such persons are believed to be at approximately 3-fold increased risk of AD dementia. We expected a majority of them to show evidence of progressive pre-clinical AD. Participants were randomized 1:1 to receive the common non-steroidal anti-inflammatory drug (NSAID) naproxen in over-the-counter dosage (naproxen sodium 220 mg) or identical-appearing placebo tablets twice daily. At baseline and at three follow-up visits (3 months, 12 months and 24 months after randomization) they were tested for cognitive abilities and undergo brain imaging with both structural and functional MRI. They are also tested for sensori-neural capacities in olfactory identification and in the ability to discern spoken language in a distracting environment (to test central auditory processing). About 2/3 of participants also volunteered to undergo a series of lumbar punctures for donation of cerebrospinal fluid (CSF), which was assayed for several biochemical markers of AD that are now understood to be present for a decade or longer before the onset of symptoms. As well, their plasma and CSF are assayed for presence of naproxen and for numerous markers of inflammatory processes (cytokines and chemokines). The central hypothesis was that administration of naproxen would not only suppress these inflammatory markers but would also slow or reverse the progress of change in cognition and in biomarkers of the pre-clinical stage of AD. The analysis plan followed the principle of modified Intent-to-Treat, considering outcomes for all persons who had at least one follow-up examination while on-protocol. After completion of two years of treatment, these participants are being followed for a further two years to observe whether treatment-related changes are sustained -- indicating that the treatment effects represent modification of the disease process itself, as opposed to a temporary change in brain function.

ELIGIBILITY:
Inclusion Criteria:

* good physical health including normal hemoglobin and hematocrit
* history or documentation of AD dementia in at least one parent, or in two siblings
* cognitive performance without diagnosable deficit such as dementia, "mild cognitive impairment"
* must have spouse or companion able to accompany participant for clinic visits
* six or more years of formal education
* fluent in either English or French
* provision of informed consent

Exclusion Criteria:

* no current peptic ulcer disease
* no history of prior peptic ulcer with bleed, perforation, intestinal obstruction
* no major psychiatric disturbance
* no regular use (4 or more doses per week) of aspirin, other non-steroidal anti-inflammatory drug (NSAID), opiate or other pain medication
* no use, present or past, of acetylcholinesterase inhibitors or memantine
* no regular use of vitamin E at dosage of 600 i.u.
* no drug or alcohol dependence
* no allergy to NSAIDs or sulfa antibiotics

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Trajectory of composite Alzheimer Progression Score (APS) from multiple cognitive and biomarker measures of pre-clinical Alzheimer's disease | Two years for primary outcome, with intent to follow participants off-treatment for two-year observational delayed washout
  Summary score derived using latent trait Item Response Theory analyses, trajectory estimated from mixed effects models based on multiple individual markers observed at baseline, three months, 12 months, and 24 months following randomization

SECONDARY OUTCOMES:
frequency and severity of treatment-emergent adverse events | collected in real-time over two years following RZ
  classified by organ system involvement and need for treatment interruption or cessation.
trajectory of cognitive abilities measured by global score on Repeatable Battery for Assessment of Neuropsychological Status | observed at baseline, annually thereafter over two years following randomization (RZ), and two years further (delayed washout)
  global score of primary interest, although individual scale scores will be used in secondary analyses
ratio of total and protein-bound naproxen concentrations as well as kinetics of drug accumulation and washout | estimated at three months and annually thereafter for two years following RZ, with further two years delayed washout
  estimate of blood brain barrier permeability and rapidity of drug accumulation and washout in both plasma and CSF partitions
biomarkers of inflammatory processes | measured at three months and annually thereafter for two years following RZ, with further two years delayed washout
  quantitative measures of 44 different inflammatory cytokines measured in plasma, and in CSF when available
CSF biomarkers of AD pathogenesis | observed at baseline, after three months, and annually thereafter over two years following randomization (RZ), and two years thereafter off-treatment (delayed washout)
  concentrations of total tau protein, phosphorylated tau protein, Amyloid beta 1-40 and Amyloid beta 1-42, apolipoprotein E

CONTACTS AND LOCATIONS:
Overall Officials: John C S Breitner, MD, MPH, Principal Investigator — Dept of Psychiatry, McGill University Faculty of Medicine
Locations (1):
- Douglas Hospital Research Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be made available, after completion of trial including delayed washout phase.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available for completed trial in March, 2018. Data for delayed washout / continuation phase will be made available at biennial intervals thereafter
Access Criteria: Qualified personnel should contact principal investigator and Study Coordinator for Data Sharing Agreement form, which must be completed and reviewed prior to release of data.